CLINICAL TRIAL: NCT02466386
Title: A Phase 3, Open-label, Multicenter, 12-Month Safety and Tolerability Study of SPD489 in Preschool Children Aged 4-5 Years Diagnosed With Attention-deficit / Hyperactivity Disorder
Brief Title: Safety and Tolerability Study of SPD489 in Preschool Children Aged 4-5 Years, Diagnosed With Attention-deficit/Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD489-348
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPD489 (Experimental): Participants will receive 5 milligrams (mg) of SPD489 capsule orally once daily in the morning and titrated in a step-wise fashion up to either 10 mg, 15 mg, 20 mg, or 30 mg until an optimal dose was reached within 52 weeks.
  Interventions: Drug: SPD489

INTERVENTIONS:
Drug: SPD489 — Participants will receive 5 mg of SPD489 capsule orally once daily in the morning and titrated in a step-wise fashion up to either 10 mg, 15 mg, 20 mg, or 30 mg until an optimal dose was reached.
  Other Names: Lisdexamfetamine dimesylate

SUMMARY:
The purpose of this study is to evaluate the long-term safety of SPD489 administered as a daily morning dose (5, 10, 15, 20, and 30 mg/day) in preschool children diagnosed with Attention-deficit/Hyperactivity Disorder (ADHD).

DETAILED DESCRIPTION:
This study is a long-term, open-label study where participants who participated in an antecedent SPD489 study (SPD489-211 [NCT02402166] or SPD489-347 [NCT03260205]) or through direct enrollment. Participants entering into this study will be classified as either a roll-over participants or a direct-enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is male or female aged 4-5 years inclusive at the time of consent from antecedent studies SPD489-211 or SPD489-347 or at the time of consent if directly enrolled.
2. Before completing any study-related procedures, participant's parent(s) or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the participant indicating that the participant is aware of the investigational nature of the study. The participant's parent(s) or LAR should understand that the required procedures and restrictions are being conducted in accordance with the International Council of Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 (1996), any updates or revisions, and applicable federal or local regulations.
3. Participant and parent(s)/LAR are willing and able to comply with all of the testing and requirements defined in the protocol, including oversight of morning dosing. Specifically, the parent/LAR should be available at approximately 7:00AM (+2 hours) to dispense the dose of investigational product for the duration of the study.
4. Roll-over participant from antecedent SPD489-347 study:

   a. Participant completed the antecedent study (SPD489-347)
5. Direct enrolled participants must meet antecedent study inclusion criteria, as listed below

   1. Participant must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV-TR) criteria for a primary diagnosis of ADHD (any subtype) based on a detailed psychiatric evaluation conducted by a sponsor-approved clinician
   2. Participant has an attention-deficit/hyperactivity disorder rating scale- IV (ADHD-RS-IV) Preschool Version total score at the Baseline Visit (Visit 0) of greater than equals to (>=) 28 for boys and >= 24 for girls.
   3. Participant has a Clinical Global Impressions - Severity of Illness (CGI-S) score >=4 at the Baseline Visit (Visit 0).
   4. Participant has a Peabody Picture Vocabulary Test, Fourth Edition standard score of >=70 at the Screening Visit (Visit -1).
   5. Participant has undergone an adequate course of non-pharmacological treatment based on investigator judgment or the participant has a severe enough condition to consider enrollment without undergoing prior non-pharmacological treatment, based on investigator judgment.
   6. Participant has, in the opinion of the investigator, participated in a structured group activity (eg, preschool, sports, Sunday school) so as to assess symptoms and impairment in a setting outside the home.
   7. Participant has lived with the same parent(s) or guardian for >=6 months.

Exclusion Criteria:

1. Participant was terminated from an antecedent SPD489 study for non-compliance and/or experienced a serious adverse event (SAE) or adverse event (AE) resulting in termination.
2. Participant is required to or anticipates the need to take medications that have central nervous system effects or affect performance, such as, but not limited to, sedating antihistamines and decongestant sympathomimetics, or monoamine oxidase inhibitors. Stable use of bronchodilator inhalers is not exclusionary.
3. Participant has a concurrent chronic or acute illness (such as, but not limited to, severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the participant. Similarly, the participant will be excluded if he or she has any additional condition(s) that, in the investigator's opinion, would prohibit the participant from completing the study or would not be in the best interest of the participant. The additional condition(s) would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. Mild, stable asthma is not exclusionary.
4. Participant has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
5. Participant has a known family history of sudden cardiac death or ventricular arrhythmia.
6. Participant has a blood pressure measurement >= 95th percentile for age, sex, and height at the screening visit (Visit -1) or the baseline visit (Visit 0) or a history of moderate or severe hypertension.
7. Participant has a known history of symptomatic cardiovascular disease, unexplained syncope, exertional chest pain, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems placing them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
8. Participant is taking any medication that is excluded per the protocol.
9. Participant had any clinically significant electrocardiogram (ECG) or clinical laboratory abnormalities at the Screening Visit (Visit -1) or baseline visit (Visit 0), based on investigator judgment.
10. Participant has a history of hyperthyroidism, or current abnormal thyroid function, defined as abnormal thyroid stimulating hormone (TSH) and thyroxine (T4) at the Screening Visit (Visit-1) or Visit 0. Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
11. Participant has taken another investigational product or has taken part in a clinical study within 30 days prior to the Screening Visit (Visit -1).
12. Participant is well-controlled on his/her current ADHD medication with acceptable tolerability.
13. Participant has glaucoma.
14. Participant has failed to fully respond, based on investigator judgment, to an adequate course of amphetamine therapy.
15. Participant has a current, controlled (requiring medication or therapy) or uncontrolled, comorbid psychiatric disorder including but not limited to any of the below co-morbid Axis I disorders and Axis II disorders:

    1. post-traumatic stress disorder (PTSD) or adjustment disorder
    2. bipolar illness, psychosis, or family history of these disorders
    3. pervasive developmental disorder
    4. obsessive-compulsive disorder (OCD)
    5. psychosis/schizophrenia
    6. participant has a serious tic disorder, or a family history of Tourette's disorder
    7. participant is currently considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation. Participants with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the investigator
    8. a history of physical, sexual, or emotional abuse
    9. any other disorder or agitated state that in the opinion of the investigator, contraindicates SPD489 or lisdexamfetamine dimesylate treatment or confound efficacy or safety assessments.
16. Participant has initiated behavioral therapy within 1 month of the baseline visit (Visit 0). Participant may not initiate behavioral therapy during the study.
17. Participant has a height <=5th percentile for age and sex at the screening visit (Visit -1).
18. Participant has a weight <=5th percentile for age and sex at the screening visit (Visit -1).
19. Participant lives with anyone who currently abuses stimulants or cocaine.
20. Participant has a history of seizures (other than infantile febrile seizures).

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shire Physician, Study Director — Shire
Locations (50):
- United States (50):
  - Harmonex, Inc, Dothan, Alabama
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Sun Valley Research Center, Imperial, California
  - Alliance for Wellness d/b/a Alliance for Research, Long Beach, California
  - AVIDA, Newport Beach, California
  - Asclepes Research, Panorama City, California
  - Psychiatric Centers at San Diego, San Diego, California
  - University of California, San Francisco, California
  - Elite Clinical Trials, Inc, Wildomar, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - APG Research, LLC, Orlando, Florida
  - University of South Florida, St. Petersburg, Florida
  - University of South Florida Department Of Psychiatry, Tampa, Florida
  - iResearch Atlanta LLC, Decatur, Georgia
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Clinical Neurophysiology Services, Sterling Heights, Michigan
  - Washington University, St Louis, Missouri
  - Premier Psychiatric Reseach Institute, LLC, Lincoln, Nebraska
  - Center For Psychiatry and Behavioral Medicine In, Las Vegas, Nevada
  - Jersey Shore University Medical Center (JSUMC), Neptune City, New Jersey
  - Manhattan Behavioral Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Duke Child and Family Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Cyn3rgy Research Center, Gresham, Oregon
  - Rainbow Research Inc, Barnwell, South Carolina
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - BioBehavioral Research of Austin, Austin, Texas
  - Bayou City Research Limited, Houston, Texas
  - BI Research Center, Houston, Texas
  - Red Oak Psychiatry Associates, Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Ericksen Research and Development, Clinton, Utah
  - Clinical Research Partners, LLC, Petersburg, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Seattle Childrens Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Childress AC, Lloyd E, Johnson SA Jr, Gunawardhana L, Arnold V. A Long-Term, Open-Label Safety and Tolerability Study of Lisdexamfetamine Dimesylate in Children Aged 4-5 Years with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2022 Mar;32(2):98-106. doi: 10.1089/cap.2021.0138. Epub 2022 Mar 8. PMID 35230142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 32 sites in United States of America from 21 August 2015 (first participant first visit) to 03 January 2020 (last participant last visit).
Pre-assignment Details: A total of 113 participants were enrolled and received the treatment. Out of which 69 participants completed the study. Since information from antecedent studies was exploratory in nature and was not really pivotal to the key conclusions of this study, only overall participant data was planned, analyzed and reported to avoid double-counting.
Groups:
- SPD489: Participants received 5 milligrams (mg) of SPD489 capsule orally once daily in the morning and titrated in a step-wise fashion up to either 10 mg, 15 mg, 20 mg, or 30 mg until an optimal dose was reached within 52 weeks.
Period: Overall Study
Arm/Group | SPD489
Started | 113
Completed | 69
Not Completed | 44
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 5
Not completed — Lack of Efficacy | 8
Not completed — Other | 10

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all participants who took at least 1 dose of investigational product.
Arm/Group | SPD489
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.8 (0.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 42
  White | 63
  More than one race | 2
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs was defined as AEs that start or deteriorate on or after the date of the first dose of investigational product and no later than 3 days following the last dose of investigational product.
Time Frame: From start of study drug administration up to follow-up (Week 53)
Population: Safety analysis set consisted of all participants who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 113
Participants | 86

2. Primary Outcome: Change From Baseline in Sleep Patterns Assessed by Children's Sleep Habits Questionnaire (CSHQ) at Week 52/ Early Termination (ET)
Description: Sleep patterns included sleep diary data and children's sleep habits questionnaire (CSHQ), which was parent report questionnaire designed to screen for the most common sleep problems in children, and consisted of 33 items for scoring and several extra items intended to provide administrators with other potentially useful information about respondents. The instrument evaluates the child's sleep based on behavior within 8 different sub scales: bedtime resistance, sleep-onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep-disordered breathing, and daytime sleepiness. Each item receives a score from 1 (problem occurs rarely) to 3 (problem usually occurs); therefore, a higher score is the worse outcome. Scale ranges are as follows: bedtime resistance: 6 to 18, sleep onset delay: 1 to 3, sleep duration: 3 to 9, sleep anxiety: 4 to 12, night walkings: 3 to 9, parasomnias: 7 to 21, sleep-disordered breathing: 3 to 9, and daytime sleepiness: 8 to 24.
Time Frame: Week 52/ET
Population: Safety analysis set consisted of all participants who took at least 1 dose of investigational product. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure at the specific categories.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | SPD489
Number analyzed (Participants) | 102
Score on scale
  Bedtime Resistance: Week 52/ET | 8.9 (3.04)
  Sleep-onset Delay: Week 52/ET | 1.6 (0.67)
  Sleep Duration: Week 52/ET | 3.8 (1.26)
  Sleep Anxiety: Week 52/ET: number analyzed (Participants) | 101
  Sleep Anxiety: Week 52/ET | 5.5 (2.09)
  Night Wakings: Week 52/ET | 4.2 (1.59)
  Parasomnias: Week 52/ET: number analyzed (Participants) | 99
  Parasomnias: Week 52/ET | 8.6 (1.54)
  Sleep-disordered Breathing: Week 52/ET | 3.4 (0.74)
  Daytime Sleepiness: Week 52/ET | 10.1 (3.78)

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Changes in Electrocardiogram (ECG) Parameters at Week 52/ Early Termination (ET)
Description: 12-lead ECG was evaluated and recorded. ECG variables included heart rate, PR interval, QRS interval, QT interval, and corrected QT interval (QTc). The QTc was calculated using both Bazett (QTcB=QT/[RR]1/2) and Fridericia (QTcF=QT/[RR]1/3) corrections. Here, > = represents "greater than or equal to", < represents "lesser than" and > represents "greater than".
Time Frame: Week 52/ET
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 99
Participants
  Heart Rate (< 55 Beats per minute) | 0
  Heart Rate (> 130 Beats per minute) | 0
  PR Interval (>= 200 millisecond [msec]) | 0
  QRS Interval (>= 90 msec) | 3
  QT Interval (> = 440 msec) | 0
  QTcB Interval (> = 440 msec and < 480 msec) | 5
  QTcB Interval (>= 480 msec and < 500 msec) | 0
  QTcB Interval (>= 500 msec) | 0
  QTcF Interval (> = 440 msec and < 480 msec) | 0
  QTcF Interval (>= 480 msec and < 500 msec) | 0
  QTcF Interval (>= 500 msec) | 0
  ECG Interpretation | 0
  ECG Abnormality - Rhythm: number analyzed (Participants) | 6
  ECG Abnormality - Rhythm | 0

4. Primary Outcome: Number of Participants With a Positive Response Using Columbia Suicide Severity Rating Scale (C-SSRS) at Week 52/ Early Termination (ET)
Description: C-SSRS was semi-structured interview that captured the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview included definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred. The C-SSRS contained 2 required items pertaining to suicidal ideation, 4 required items pertaining to suicidal behavior, and 1 required item pertaining to non-suicidal but self-injurious behavior. In situations where there was a positive response to the screening questions, there were 8 additional suicidal ideation items and 4 additional suicidal behavior items which were completed. Thus, there was a maximum of 19 items to be completed. Here number of participants responded as yes to suicidal ideation or behaviour were reported.
Time Frame: Week 52/ET
Population: Safety analysis set consisted of all participants who took at least 1 dose of investigational product. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 112
Participants | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Changes in Clinical Laboratory Values at Week 52/ Early Termination (ET)
Description: Clinical laboratory evaluations included biochemistry and endocrinology, hematology, and urinalysis. Number of participants with potentially clinically significant changes in clinical laboratory values were reported.
Time Frame: Week 52/ET
Population: Safety analysis set consisted of all participants who took at least 1 dose of investigational product. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure and at the specific categories.
Measure: Count of Participants; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 104
Participants
  Hematology: Eosinophils/Leukocytes: Greater than (>)10% | 12
  Hematology: Hematocrit: Less than (<) 0.3 | 2
  Hematology: Leukocytes: <3 × 10^9/Liter (L) | 1
  Hematology: Leukocytes: >16 × 10^9/L | 1
  Hematology: Lymphocytes/leukocytes: >70% | 1
  Hematology: Neutrophils: <1 × 10^9/L | 1
  Hematology: Neutrophils/leukocytes: <30% | 15
  Hematology: Platelets: <75 × 10^9/L: number analyzed (Participants) | 103
  Hematology: Platelets: <75 × 10^9/L | 1
  Biochemistry and Endocrinology: Glucose: <3.05 Millimole per liter (mmol/L) | 2
  Biochemistry and Endocrinology: Glucose: >8.88 mmol/L | 2
  Biochemistry and Endocrinology: Potassium: >5.5 mmol/L | 1
  Biochemistry and Endocrinology: Protein: >90 gram per liter (g/L) | 1
  Biochemistry and Endocrinology: Thyrotropin: < Lower limit of normal (LLN): number analyzed (Participants) | 103
  Biochemistry and Endocrinology: Thyrotropin: < Lower limit of normal (LLN) | 7
  Urinalysis: Ketones: Positive value (excluding trace): number analyzed (Participants) | 103
  Urinalysis: Ketones: Positive value (excluding trace) | 15
  Urinalysis: Occult blood: Positive value (excluding trace): number analyzed (Participants) | 103
  Urinalysis: Occult blood: Positive value (excluding trace) | 2
  Urinalysis: Protein: Positive value (excluding trace): number analyzed (Participants) | 103
  Urinalysis: Protein: Positive value (excluding trace) | 30

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Changes in Vital Signs at Week 52/ Early Termination (ET)
Description: Vital sign assessments included blood pressure, pulse and respiratory rate. Number of participants with potentially clinically significant changes in vital signs were reported.
Time Frame: Week 52/ET
Population: Safety analysis set consisted of all participants who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 113
Participants | 0

7. Secondary Outcome: Clinical Global Impressions Global Improvement (CGI-I) at Week 52/ Early Termination (ET)
Description: CGI-I was an overall assessment of global symptom improvement by evaluation of the participant's condition severity and improvement over time. Scoring was done based on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), where higher score reported worse condition. The scoring was elaborated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Week 52/ET
Population: Full analysis set consisted of all participants in the safety analysis set who took at least 1 post-dose ADHD-RS-IV Preschool Version Total Score assessment during the study. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SPD489
Number analyzed (Participants) | 87
Score on a scale | 2.0 (0.91)

8. Secondary Outcome: Change From Baseline in Clinician-Administered Attention-Deficit/Hyperactivity Disorder Rating Scale-IV (ADHD-RS-IV) Preschool Version Total Score at Week 52/ Early Termination (ET)
Description: ADHD-RS-IV Preschool Version was adapted from the ADHD Rating Scale-IV and provided examples appropriate for the developmental level of preschool children. The ADHD-RS-IV Preschool Version was an 18-item questionnaire that required the respondent to rate the frequency of occurrence of ADHD symptoms as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition-Text Revision (DSM-IV-TR) criteria. Each item was scored on a 4-point scale ranging from 0 (never or rarely) to 3 (very often) with total scores ranging from 0-54. The 18 items were grouped into 2 subscales: hyperactivity/impulsivity (even numbered items 2-18) and inattentiveness (odd numbered items 1-17).
Time Frame: Week 52/ET
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SPD489
Number analyzed (Participants) | 87
Score on a scale | -24.2 (13.34)

9. Primary Outcome: Number of Participants With Shift From Baseline in Body Mass Index (BMI) Percentiles at Week 52/Early Termination (ET)
Description: BMI was derived from height and weight. BMI was normalized by sex and age using the CDC growth charts. BMI percentiles were categorized as: Underweight (BMI < 5th percentile); Healthy weight (BMI 5th percentile up to < 85th percentile); Overweight (BMI 85th percentile < 95th percentile); Obese (BMI >= 95th percentile). Number of participants with shift from baseline in BMI percentile categories at Week 52/ET was reported.
Time Frame: Week 52/ET
Population: Safety analysis set consisted of all participants who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 113
Participants
  Underweight: Week 52/ET | 8
  Healthy Weight: Week 52/ET | 78
  Overweight: Week 52/ET | 12
  Obese: Week 52/ET | 3

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Week 53)
Groups:
- Total: Participants received 5 mg of SPD489 capsule orally once daily in the morning and titrated in a step-wise fashion up to either 10 mg, 15 mg, 20 mg, or 30 mg until an optimal dose was reached within 52 weeks.
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 0/113
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 57/113
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total (N=113)
Vomiting (Gastrointestinal disorders) | 6 (7)
Pyrexia (General disorders) | 11 (12)
Influenza (Infections and infestations) | 10 (10)
Nasopharyngitis (Infections and infestations) | 8 (11)
Pharyngitis streptococcal (Infections and infestations) | 9 (11)
Upper respiratory tract infection (Infections and infestations) | 8 (15)
Weight decreased (Investigations) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 18 (21)
Affect lability (Psychiatric disorders) | 7 (8)
Initial insomnia (Psychiatric disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (4):
  • Study Protocol: Protocol (2014-10-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT02466386/Prot_000.pdf
  • Study Protocol: Amendment 1 (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT02466386/Prot_001.pdf
  • Study Protocol: Amendment 2 (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT02466386/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT02466386/SAP_003.pdf